CLINICAL TRIAL: NCT05928949
Title: Effect of Pilates Exercises on Balance and Gross Motor Co-Ordination In Children With Down Syndrome
Brief Title: Pilates Exercises and Down Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Fahmy Hassan Al Nemr, PHD, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: P.T.REC/012/003399
Record Dates: First submitted 2023-06-25; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-01

CONDITIONS: Balance; Down Syndrome; Pilates Exercises
MeSH Terms: conditions — Down Syndrome | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy (Active Comparator): Group A performed flexibility, strength, and endurance exercises that focused on the lower extremity and trunk muscles, exercise for postural stability in various positions and surfaces, including flexibility exercises for the hip, knee and calf muscle. Strengthening exercises included the core muscles, hip abductors, hip extensors hamstrings and quadriceps knee extension in high sitting. Postural control involved walking in all directions, exceeding the limits of stability in various positions such as kneeling, half kneeling, standing on rough and soft surfaces, Each session started with a warming up and cooling down of 5 minutes for each period and each session lasted for 45 minutes.
  Interventions: Other: pilates exercises
- pilates exercises (Experimental): group B received the same program of exercises given to group A in addition to 45 minutes of Pilates exercises to improve balance and gross motor coordination. Exercises were performed on a mat, a medical ball, and from a standing position, focusing on maintaining core contraction, spinal and pelvic alignment, and respiration rhythm. Ten repetitions of Pilates exercises will be performed with a 2-minute rest period between repetitions. Both groups will attend the intervention program three times/week for 3 months
  Interventions: Other: pilates exercises

INTERVENTIONS:
Other: pilates exercises — Pilates is a system of repetitive exercises performed on a yoga mat or other equipment to promote strength, stability, and flexibility. Pilates exercises develop the body through muscular effort that stems from the core.

SUMMARY:
Down syndrome is one of the genetic disorders that affect postural control and balance in children. Balance involves controlling the position of the body in space to achieve stability and orientation. pilates exercises are one of several techniques that are used to improve balance and postural control in adults and children.

the purpose of the study is To investigate the effect of Pilates exercises on balance and gross motor co-ordination in children with Down syndrome

DETAILED DESCRIPTION:
Group A performed flexibility, strength, and endurance exercises that focused on the lower extremity and trunk muscles, exercise for postural stability in various positions and surfaces, including flexibility exercises for the hip, knee and calf muscle. Strengthening exercises included the core muscles, hip abductors, hip extensors hamstrings and quadriceps knee extension in high sitting. Postural control involved walking in all directions, exceeding the limits of stability in various positions such as kneeling, half kneeling, standing on rough and soft surfaces, Each session started with a warming up and cooling down of 5 minutes for each period and each session lasted for 45 minutes.

Group B received the same program of exercises given to group A in addition to 45 minutes of Pilates exercises to improve balance and gross motor coordination. Exercises were performed on a mat, a medical ball, and from a standing position, focusing on maintaining core contraction, spinal and pelvic alignment, and respiration rhythm. Ten repetitions of Pilates exercises will be performed with a 2-minute rest period between repetitions. Both groups will attended the intervention program three times/week for 3 months

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosed with Trisomy 21 through genetic testing, (2) aged 6 to 11 years and (3) able to follow a minimum of two-step instructions. The minimum motor ability of participants with DS was independent locomotion.

Exclusion Criteria:

* (1) medical condition that is contraindicated to moderate to vigorous physical activity such as cardiovascular problems, (2) orthopaedic instability, including those associated with DS (e.g. atlanto-axial instability) and (3) behavioural issues that hindered instruction.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-06-26 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-11 (Estimated)

PRIMARY OUTCOMES:
balance | 3 months
  Balance assessment will be performed in both groups before and after the intervention to find any significant difference, by using the Biodex Balance System to evaluate all measurable variables of stability indices (anteroposterior stability index and mediolateral stability index).
Bruininks-oseretsky test of motor proficiency-second version (BOT-2) | 3 months
  BOT-2 measures gross motor proficiency, with subtests that focus on stability, mobility, strength, coordination, and object manipulation. The test is tailored to school-aged children, who have varying motor control abilities ranging from normal to mild or moderate. In this study, it will be used to measure gross motor co-ordination.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Physical Therapy, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Nemr A, Reffat S. Effect of Pilates exercises on balance and gross motor coordination in children with Down syndrome. Acta Neurol Belg. 2024 Oct;124(5):1499-1505. doi: 10.1007/s13760-024-02517-w. Epub 2024 Apr 1. PMID 38558387